CLINICAL TRIAL: NCT07248410
Title: A Split-Scalp Study Evaluating the Efficacy and Safety of Fractional Laser Therapy With and Without Exosomes in the Treatment of Androgenetic Alopecia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: ExoOne bio (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ExoOne-CS-2025001a
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Androgenetic Alopecia
Keywords: Androgenetic Alopecia; exosome; minoxidil; fractional laser
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A: left scalp: exosome/right scalp: normal saline (Other): During the first 3 months, participants received fractional laser treatment once a month. The left scalp was applied with exosome product once in the morning and once in the evening, while the right scalp was applied with normal saline once in the morning and once in the evening, with each dose being 1 ml. During the next 3 months, the left scalp was applied with the exosome product once in the morning and once in the evening, while the right scalp was applied with normal saline once in the morning and once in the evening.
  Interventions: Device: fraction laser
- B: right scalp: exosome/left scalp: normal saline (Other): During the first 3 months, participants received fractional laser treatment once a month. The right scalp was applied with exosome product once in the morning and once in the evening, while the left scalp was applied with normal saline once in the morning and once in the evening, with each dose being 1 ml. During the next 3 months, the right scalp was applied with the exosome product once in the morning and once in the evening, while the left scalp was applied with normal saline once in the morning and once in the evening.
  Interventions: Device: fraction laser

INTERVENTIONS:
Device: fraction laser — We will performed the fraction laser on the scalp of participants with energy of 30-40mJ every month for 3 times.

SUMMARY:
This trial aims to evaluate the efficacy, safety, and tolerability of fractional laser combined with topical exosome for hair regrowth in patients with androgenetic alopecia.

This study is expected to recruit 30 participants. The experimental group will receive fractional laser treatment combined with human umbilical cord mesenchymal stem cell exosome solution; the control group will receive fractional laser treatment combined with a placebo. Participants will receive three fractional laser treatments and will be followed up for 6 months. At each follow-up visit, hair density, diameter, vellus hair to terminal hair ratio, and adverse reactions will be assessed using trichotomy; a global photographic assessment will be performed using standardized imaging equipment.

ELIGIBILITY:
Inclusion Criteria:

1. Male pattern baldness diagnosed according to the Norwood-Hamilton classification III-V
2. Males aged 18 to 50 years
3. Willing to provide written informed consent and possessing the ability to read, write, speak, and understand
4. Able to follow the study's treatment guidelines

Exclusion Criteria:

1. Those who have taken oral Finasteride, Dutasteride, or Minoxidil within 6 months prior to the start of the trial.
2. Those who have used any topical or systemic medications that may affect hair growth within 6 months prior to the start of the trial.
3. Those who have received phototherapy, laser therapy, exosome therapy, or hair regrowth injections (such as minimally invasive procedures) within 6 months prior to the start of the trial.
4. Those with a history of hair transplant surgery.
5. Those suffering from other systemic or scalp diseases that may affect hair growth (e.g., iron deficiency anemia, immune disorders, thyroid diseases, and syphilis).
6. Those with a history of severe inflammation, keloids, malignant tumors, or poor wound healing at the treatment site.
7. Those with other diseases that make them unsuitable for fractional laser treatment.
8. Those with a history of malignant tumors or currently undergoing treatment.
9. Participants must not undergo any cosmetic procedures that may affect scalp condition or hair growth throughout the entire trial period, including hair dyeing, perming, bleaching, scalp exfoliation, deep scalp cleansing, or any other actions that may irritate or damage the scalp.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-24 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in hair density (d84) | Baseline to Day 84
  Evaluation of the change in hair density of fractional laser combined with exosomes in improving hair growth

SECONDARY OUTCOMES:
Change in hair density (d168) | Baseline to Day 168
  Evaluation of the change in hair density of fractional laser combined with exosomes in improving hair growth.
Change in Hair diameter (d168) | Baseline to Day 168
  Evaluation of the change in hair diameter of fractional laser combined with exosomes in improving hair growth.
Change in the percentage of vellus hair and terminal hair (d168) | Baseline to Day 168
  Evaluation of the change in the percentage of vellus hair and terminal hair of fractional laser combined with exosomes in improving hair growth
Change in global photographic assessment (d168) | Baseline to Day 168
  Evaluation of the change in global photographic assessment of fractional laser combined with exosomes in improving hair growth

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital Taoyuan branch, Taoyuan District, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Suchonwanit P, Rojhirunsakool S, Khunkhet S. A randomized, investigator-blinded, controlled, split-scalp study of the efficacy and safety of a 1550-nm fractional erbium-glass laser, used in combination with topical 5% minoxidil versus 5% minoxidil alone, for the treatment of androgenetic alopecia. Lasers Med Sci. 2019 Dec;34(9):1857-1864. doi: 10.1007/s10103-019-02783-8. Epub 2019 Apr 13. PMID 30982177
- [Background] Amini F, Teh JJ, Tan CK, Tan ESS, Ng ESC. A Pilot Randomized Controlled Trial (RCT) Evaluating the Efficacy of an Exosome-Containing Plant Extract Formulation for Treating Male Alopecia. Life (Basel). 2025 Mar 20;15(3):500. doi: 10.3390/life15030500. PMID 40141845
- [Background] Chen YC, Tsai WC, Li ZX, Lin WJ, Lin HY, Hsieh YJ, Wang KH, Chen YY, Hwang TL, Lin TY. Exosomes from human umbilical cord mesenchymal stem cells promote the growth of human hair dermal papilla cells. PLoS One. 2025 Apr 30;20(4):e0320154. doi: 10.1371/journal.pone.0320154. eCollection 2025. PMID 40305498